CLINICAL TRIAL: NCT00003772
Title: An International Field Study of the Reliability and Validity of a Disease-Specific Questionnaire Module (the QLQ-OV28) in Assessing the Quality of Life of Patients With Ovarian Cancer
Brief Title: Quality-of-Life Assessment in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-15982; EORTC-15982 (Other: EORTC)
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Quality-of-life assessment in patients undergoing cancer treatment may help determine the intermediate- and long-term effects of treatment.

PURPOSE: This clinical trial studies the quality of life in patients with ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the scale structure and reliability of the ovarian cancer specific questionnaire module (EORTC QLQ-OV28) designed to be used in conjunction with the standard nonspecific questionnaire (EORTC QLQ-C30) in patients with ovarian epithelial cancer. II. Evaluate the psychometric properties of the revised scales (physical and role functioning; global health status/QL) of the EORTC QLQ-C30 among ovarian cancer patients. III. Evaluate the evidence for the validity of EORTC QLQ-OV28.

OUTLINE: This is a multicenter study. Patients are stratified according to prior therapy and disease. Questionnaires are designed to be completed by patients themselves without help. Patients complete the EORTC QLQ-C30, QLQ-OV28, and a debriefing questionnaire regarding time to completion and patient's reaction to the quality of life questionnaires according to one of the following schedules: Group 1: Patients complete the questionnaires once prior to the start of the first course of chemotherapy, and again on the first day of the third course of chemotherapy. Group 2: Patients complete the questionnaires once 1 to 8 weeks following completion of the 6th course of chemotherapy and prior to any further anticancer therapy. Group 3: Patients complete the questionnaires once at a routine follow-up clinic visit and again at home within 3 days of the clinic visit. Group 4: Patients complete the questionnaires once prior to the first course of chemotherapy and again on the first day of the 3rd course of chemotherapy prior to administration OR at the first clinical review following 2 courses of chemotherapy OR 2 months later for patients receiving continuous or weekly chemotherapy. If they are unable to complete written questionnaires due to physical limitations or illiteracy, or if they express a strong preference for oral administration, patients in Groups 1, 2, and 4 may complete the questionnaires orally instead.

PROJECTED ACCRUAL: A minimum of 280 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of ovarian epithelial carcinoma No prior participation in this study as a member of a different group Group 1: Prior surgery required Scheduled for first line chemotherapy No chemotherapy prior to surgery Group 2: Prior surgery required Completion of 6 courses of first line platinum-based chemotherapy required within 8 weeks prior to study Group 3: Must have achieved complete response to first line therapy At least 3 months since any therapy for cancer Prior surgery required Prior chemotherapy allowed Prior radiotherapy allowed Group 4: Must have recurrent disease Scheduled for chemotherapy Prior surgery required Prior chemotherapy allowed Prior radiotherapy allowed

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No concurrent malignancies except basal cell carcinoma of the skin No mental disease or language barrier that would prevent compliance No concurrent participation in any other quality of life study that might interfere with this study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 1999-01; Primary Completion 2001-08 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cull, PhD, Study Chair — Edinburgh Cancer Centre at Western General Hospital
Locations (4):
- Landeskrankenhaus/Universitatskliniken Graz, Graz, Austria
- Centre Alexis Vautrin, Vandœuvre-lès-Nancy, France
- Hospital De Navarra, Pamplona, Spain
- Western General Hospital, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Result] Chie WC, Tsai CJ, Chiang C, Lee YC. Quality of life of patients with oesophageal cancer in Taiwan: validation and application of the Taiwan Chinese (Mandarin) version of the EORTC QLQ-OES18: a brief communication. Qual Life Res. 2010 Oct;19(8):1127-31. doi: 10.1007/s11136-010-9675-8. Epub 2010 May 22. PMID 20495876
- [Result] Cull A, Howat S, Greimel E, Waldenstrom AC, Arraras J, Kudelka A, Chauvenet L, Gould A; EORTC Quality of Life Group [European Organization for Research and Treatment of Cancer]; Scottish Gynaecological Cancer Trials Group. Development of a European Organization for Research and Treatment of Cancer questionnaire module to assess the quality of life of ovarian cancer patients in clinical trials: a progress report. Eur J Cancer. 2001 Jan;37(1):47-53. doi: 10.1016/s0959-8049(00)00369-5. PMID 11165129